CLINICAL TRIAL: NCT05691322
Title: Prospective Validation of the DEVA Algorithm for the Prediction of Severe Endometriosis
Acronym: ValDEVA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: One Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: ValDEVA-01
Record Dates: First submitted 2023-01-06; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: transvaginal ultrasound — Transvaginal ultrasound for endometriosis diagnosis (UBESS)
Diagnostic Test: MRI — MRI for endometriosis diagnosis (Enzian classification)

SUMMARY:
Endometriosis is a chronic disease affecting 1 in 10 women. Its diagnosis is difficult and the time between the first symptoms and diagnosis is of about 7 years. diagnosis requires specialized imaging performed by referral practitioners for this pathology. According to current recommendations, non-specialized pelvic ultrasound is the recommended first-line examination. However, only reference ultrasound, performed by a doctor specialized in the disease and carried out according to a specific protocol (such as UBESS), is sufficiently reliable for diagnosis. The number of practitioners performing this type of examination is very low in France, which in practice results in a very low reliability of this strategy in real life. Pelvic MRI is also a much more reliable examination, available for review. However its access is limited. In addition, the false positive rate can be as high as 20%, particularly for minor forms of the disease.

The DEVA algorithm has been developed for the identification of women with endometriosis based on a self-administered pelvic pain symptom questionnaire (ENDOPAIN). In a preliminary study, this algorithm seems reliable for identify patients at high risk of this disease and would thus allow to triage patients requiring patients requiring an immediate MRI in order to shorten diagnostic delays. External validation of the algorithm is therefore necessary before clinical use. The main objective od this study is the prospective external validation of the diagnostic reliability of the DEVA algorithm used for the detection of women with endometriosis (visible on MRI or transvaginal ultrasound).

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* patients aged 18-45
* Patients addressed for an pelvic IRM or transvaginal echography

Exclusion Criteria:

* Minor patients
* Patients Over 45 years of age
* Patients without social security
* Patients that do not know how to read in French
* Patients with a chronic pathology responsible of pain or handicap
* Patients with a major pelvic pathology
* Patients with more than 3 months of amenorrhea
* Patients diagnosed or suspicious of having an invasive cancer.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Female volunteers aged 18-45 years, referred for pelvic MRI or transvaginal ultrasound referral regardless of symptomatology. The practitioners performing the examinations are recognised for their experience in the diagnosis of diagnosis of endometriosis.
Sampling Method: Probability Sample
Enrollment: 276 (Estimated)
Dates: Start 2022-10-19 (Actual); Primary Completion 2023-10-19 (Estimated); Study Completion 2024-01-19 (Estimated)

PRIMARY OUTCOMES:
Positive likelihood ratio of the algorithm classification based on the MRI or UBESS US results | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Intercommunal Poissy Saint Germain, Poissy, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fauconnier A, Drioueche H, Huchon C, Du Cheyron J, Indersie E, Candau Y, Panel P, Fritel X. Early identification of women with endometriosis by means of a simple patient-completed questionnaire screening tool: a diagnostic study. Fertil Steril. 2021 Dec;116(6):1580-1589. doi: 10.1016/j.fertnstert.2021.07.1205. Epub 2021 Sep 17. PMID 34538656